CLINICAL TRIAL: NCT02773264
Title: Validation of Ultra Sound (US) Elastography for the Evaluation of Soft Tissue and Organ Lesions
Brief Title: Validation of Ultra Sound (US) Elastography
Acronym: USE
Status: Terminated | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: idr-us-001
Record Dates: First submitted 2015-06-02; First posted 2016-05-16 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Soft Tissue Lesions
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- UltraSound Patients: All patients will undergo next to the clinical indicated conventional US-examination, US Elastography after informed consent. After completion of these three examinations, the participation in the study is completed.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound Elastography of soft tissue and organ lesions

SUMMARY:
This is a prospective, single-center, non-randomised, non-blinded trial with US Elastography of Patients referred to our institution to assess soft tissue and organ lesions. All patients will undergo next to the clinical indicated conventional US-examination, US Elastography after informed consent. After completion of these three examinations, the participation in the study is completed.

DETAILED DESCRIPTION:
The investigators propose UltraSound Elastography as an imaging method which allows for a better evaluation of soft tissue and organ lesions compared to the conventional US modalities used nowadays in the dayly clinical routine.

This is a prospective, single-center, non-randomised, non-blinded trial with US Elastography of Patients referred to our institution to assess soft tissue and organ lesions. All patients will undergo next to the clinical indicated conventional US-examination, US Elastography after informed consent. After completion of these three examinations, the participation in the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for clinically indicated conventional Ultrasound examination

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for clinically indicated conventional Ultrasound examination
Sampling Method: Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2016-03-01; Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Non-Inferiority to conventional Ultrasound (conv. US) | when scheduled for conv. US, 30minutes
  Value of US Elastography compared to conventional US

SECONDARY OUTCOMES:
Superiority to conventional Ultrasound (conv. US) | when scheduled for conv. US, 30minutes
  Value of US Elastography compared to conventional US

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frauenfelder, PD MD, Principal Investigator — University Hospital Zurich, Institue of Diagnostic Radiology
Locations (1):
- University Hospital Zurich - Diagnostic Radiology, Zurich, Switzerland

REFERENCES:
- See also: Elastography in pancreatic solid tumours diagnoses. — http://www.ncbi.nlm.nih.gov/pubmed/25960814